CLINICAL TRIAL: NCT00793078
Title: Investigation of Arterial Blood Pressure-complexity and Its Relation to Outcome in Comparison Between Cardiac Surgery Versus Non-cardiac Surgery Septic Patients
Brief Title: Arterial Blood Pressure-complexity in Septic Patients
Status: Suspended | Type: Observational
Why Stopped: Awaiting decision on financial support by Deutsche Forschungsgemeinschaft (DFG)
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Priv.-Doz. Dr. med. Martin Soehle, D.E.S.A., Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn
Other Study IDs: VCS2009
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-01

CONDITIONS: Sepsis
Keywords: sepsis; arterial blood pressure; complexity; variability
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Arterial blood pressure (ABP) is regulated by multiple, interconnected feedback loops resulting in a variable and complex time course. According to the "decomplexification theory of illness", disease is characterised by a loss or impaired function of feedback loops resulting in a decreased complexity of the ABP-time course and an impaired adaptability of the cardiovascular system.

Decomplexification of physiologic parameters has been shown to occur in coronary heart disease, Parkinson's and Hodgkin's disease, and in subarachnoid hemorrhage, but has not been evaluated in sepsis.

This study is intended to test the hypothesis that complexity of ABP

* is lower in cardiac surgery versus non-cardiac surgery septic patients,
* decreases as severity of sepsis increases to severe sepsis and septic shock,
* is associated with outcome three month after sepsis.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from sepsis, severe sepsis or septic shock

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated at the Intensive Care Unit of a University Hospital
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
short form-36 | 3 month after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soehle, M.D., D.E.S.A., D. habil., Principal Investigator — Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Bonn, Germany